CLINICAL TRIAL: NCT00867425
Title: Translating the Diabetes Prevention Program Into a Virtual Lifestyle Management Program: A Pilot Study in a Military Community
Brief Title: Translating the Diabetes Prevention Program Into a Virtual Lifestyle Management Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: U.S. Air Force Office of the Surgeon General (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kathleen McTigue, Assistant Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PRO08030183; FWH20080195H
Record Dates: First submitted 2009-03-20; First posted 2009-03-23 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Obesity; Diabetes; Cardiovascular Disease
Keywords: Diabetes; Internet; Obesity; Obesity with high cardiovascular risks
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental)
  Interventions: Behavioral: Virtual Lifestyle Management

INTERVENTIONS:
Behavioral: Virtual Lifestyle Management — The VLM online lifestyle intervention will include elements of a behavioral lifestyle program developed by the Diabetes Prevention Program (1). VLM will assist individual participants with establishing appropriate weight loss goals, implementing dietary recommendations (including analysis of current diet), and defining exercise programs.
  Participants will be encouraged to complete 16 online, weekly lessons. The VLM curriculum provides standard information about healthy lifestyle, and behavioral techniques for integrating them into daily living. In each lesson, patients provide feedback about how they interpret the information, and ideas for integrating it into their lives. The VLM lifestyle coaching team will review these entries weekly, and provide support, feedback about progress, tips on how to problem-solve around lifestyle barriers, and guidance on how to use the "Keeping Track" functions of VLM (e.g. keeping track of weight, fat intake, calories or physical activity).
  Other Names: Diabetes Prevention Program

SUMMARY:
The objective of this study is to evaluate the effectiveness of Virtual Lifestyle Management (VLM) as a behavior modification tool to promote weight loss, healthy eating and physical activity patterns, in the interest of reducing risk and adverse outcomes for individuals at high risk of type 2 diabetes (T2D) and cardiovascular disease (CVD) in a military population.

Specific Aim: To evaluate the effect of VLM on cardiovascular risk status in participants at high risk or individuals with T2D enrolled in the pilot study. The investigators hypothesize that participants will show greater improvement in weight as well as glucose, blood pressure, lipids, and self-reported diet and physical activity than will similar patients who are not enrolled in VLM.

DETAILED DESCRIPTION:
As the epidemic of obesity continues to grow in both the United States and military populations, innovative lifestyle interventions that fit into the schedules of a busy population are critical. The rising costs of obesity (direct medical costs as well as societal costs) are staggering, and left unaddressed, they will overwhelm the budgets of many employers. Additionally, the costs in terms of military readiness are critical. As more career soldiers choose separation over weight reduction, the loss of institutional knowledge and intellectual capital are consequences that will continue to be felt. A program that is successful, scaleable, and transferable to remote locations could help stem this tide. VLM will begin the process of allowing the internet to be used not only as an informational and communication tool, but also as a means of accessing a comprehensive and well-validated lifestyle program from the internet-access point of greatest convenience.

Type 2 diabetes (T2D) affects 18 million Americans(2) and costs $132 billion in expenditures and lost productivity.(3) Treatment and prevention are essential, yet current recommendations,(4) combining medical care with self-care, are difficult to implement. Furthermore, strong evidence supports the use of comprehensive, intensive lifestyle interventions for obesity among primary care patients. While such programs may help reduce the risk of T2D onset, assist with glucose management among individuals who have T2D, and benefit other obesity-related health problems, such programs are commonly lacking in clinical practice.

This pilot study will test a model for the implementation of a VLM program that utilizes the internet to address good nutrition, safe weight loss methods and the importance of physical activity with the "virtual" support of a lifestyle coaching team to sustain participants in their weight loss and physical activity efforts. The focus of this initiative is to promote weight loss and healthy diet and exercise patterns, in the interest of preventing and treating T2D, and minimizing the risk of CVD in the military community. The study will be open to individuals who receive medical care through Wilford Hall Medical Center (WHMC) clinics.

ELIGIBILITY:
Inclusion Criteria:

* Overweight (BMI > 25 kg/m2)
* diagnosis of at least one of the following: hypertension, dyslipidemia, type 2 diabetes, glucose intolerance
* receive health care at the 59th Medical Wing of the US Air Force
* at least weekly access to a computer with high-speed internet
* at least weekly access to a scale
* able to attend an in-person orientation session
* able to understand and sign informed consent
* agree to participate in the VLM program and evaluation

Exclusion Criteria:

* known deployment within 6 months
* Primary care physician determination that moderate physical activity and/or a low-fat diet are not safe or appropriate
* pregnancy
* breastfeeding
* current weight loss therapy
* history of bariatric surgery
* plans to have bariatric surgery

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-04; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Change in weight | 4 months

SECONDARY OUTCOMES:
Blood Pressure | 4 months
Lipids | 4 months
A1C (if applicable) | 4 months
Physical Activity | 4 months
Eating Behaviors | 4 months
Health Related Quality of Life | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M McTigue, MD, MS, MPH, Study Director — University of Pittsburgh
Locations (1):
- Wilford Hall Medical Center, Lackland Air Force Base, Texas, United States

REFERENCES:
- [Background] Diabetes Prevention Program (DPP) Research Group. The Diabetes Prevention Program (DPP): description of lifestyle intervention. Diabetes Care. 2002 Dec;25(12):2165-71. doi: 10.2337/diacare.25.12.2165. PMID 12453955
- [Background] ADA. All About Diabetes. found at http://www.diabetes.org/about-diabetes.jsp. 2004.
- [Background] Hogan P, Dall T, Nikolov P; American Diabetes Association. Economic costs of diabetes in the US in 2002. Diabetes Care. 2003 Mar;26(3):917-32. doi: 10.2337/diacare.26.3.917. PMID 12610059
- [Background] American Diabetes Association. Standards of medical care in diabetes. Diabetes Care. 2004 Jan;27 Suppl 1:S15-35. doi: 10.2337/diacare.27.2007.s15. No abstract available. PMID 14693923